CLINICAL TRIAL: NCT03079856
Title: Drug Use and Sexual Risk Behaviors Among Emerging Adults in the ER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Erin Bonar, Assistant Professor of Psychiatry, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: NIDA036008; 4K23DA036008-04 (NIH)
Record Dates: First submitted 2017-02-27; First posted 2017-03-15 (Actual); Last update posted 2018-08-29 (Actual); Status verified 2018-08

CONDITIONS: Drug Use; Sex Behavior
Keywords: Emerging adults; Drugs; HIV; Risky Sex Behaviors
MeSH Terms: conditions — Sexual Behavior | interventions — Crisis Intervention

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Brief Intervention (Experimental): ED-based computer-guided intervention for substance use and HIV risk reduction utilizing Motivational Interviewing
  Interventions: Behavioral: Brief Intervention
- Enhanced Usual Care (No Intervention): Substance use and sexual health services information within a brochure provided to participants

INTERVENTIONS:
Behavioral: Brief Intervention — Intervention for emerging adults (EAs) seeking care in the ED. The intervention will be rooted in motivational interviewing (MI) and will be guided by social cognitive, self-determination, and the trans-theoretical theories. The ED visit presents a "teachable moment" for intervening to promote health behavior, therefore eligible EAs will receive a ~30 minute MI-based session in the ED. In order to capitalize on and potentially extend this moment, participants will receive daily booster notifications delivered through a secure mobile app that they will download to their phone at enrollment.
  Arms: Brief Intervention

SUMMARY:
This project will develop a technology-augmented HIV and substance use risk reduction intervention for delivery in the Emergency Department, a medical setting where at-risk emerging adults who use drugs and engage in HIV-related risk behaviors are likely to present.

DETAILED DESCRIPTION:
Research regarding substance use (including illicit drugs and non-medical use of prescription drugs) and HIV-related sexual risk behaviors (HIV SRBs; e.g., inconsistent condom use, multiple partners, sex while intoxicated; and prevention of injection drug use) among emerging adults (EAs; ages 18-25) has generally focused on alcohol use among college students from campus settings; however, substance use and HIV (and other associated Sexually Transmitted Infections) disproportionately occur among young people living in urban, low-resource communities, particularly individuals of racial minorities. The Emergency Department (ED) is a critical venue for accessing at-risk EAs engaging in substance use and HIV risk behaviors. Research shows high rates of substance use and HIV SRBs among EA patients in the ED, yet no intervention exists for EAs in this setting. The ED may be the only opportunity to intervene with these young people because EAs in urban, low-resource settings often lack a primary care provider during the transition from pediatric to adult medicine, may be un-insured or under-insured, and may not be involved in a traditional college campus setting. Further the use of technology (e.g., mobile phones) is relatively ubiquitous among this age group, and most prefer technology-based communication (e.g., text messaging or instant messaging via apps), therefore interventions for EAs may be enhanced by this type of technology. In this phase we will test a tailored intervention for EA patients in the ED focusing on reducing substance use and HIV SRBs, which will be enhanced through the use of mobile app notifications.

ELIGIBILITY:
Inclusion Criteria:

* Medically stable
* Mentally and physically able to consent
* English-speaking
* Between ages 18-25
* Past-month substance use (including illicit drugs and/or non-medical prescription drug use) and inconsistent condom use in the past month
* Ownership of a smartphone

Exclusion Criteria:

* ED presentation suicidality and/or acute psychosis, being in police custody, or present with psychological distress requiring intensive social work (e.g. sexual assault)
* Patients with a significant other that they live with who is currently participating in study
* Actively participating in another study
* Participated in prospective and intervention development phases of the study
* Married
* Do not wish to consent to audio-taping the in-person portion of the ED-based intervention session

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 63 (Actual)
Dates: Start 2017-10-09 (Actual); Primary Completion 2018-08-13 (Actual); Study Completion 2018-08-13 (Actual)

PRIMARY OUTCOMES:
Change in days substance use | 2-months post baseline
  60-day Timeline Follow-Back (TLFB) will be used to assess total days of any substance use.
Change in quantity of marijuana use | 2-months post baseline
  60-day Timeline Follow-Back (TLFB) will be used to assess quantity of marijuana consumed.
Change in total alcohol consumption | 2-months post baseline
  60-day Timeline Follow-Back (TLFB) will be used to assess quantity of alcohol consumed

SECONDARY OUTCOMES:
Change in HIV risk behaviors | 2-months post baseline
  60-day Timeline Follow-Back (TLFB) will be used to assess frequency of unprotected sex.
Change in substance use consequences | 2-months post baseline
  Modified Rutgers Alcohol Problems Index adapted for alcohol and drugs will assess total substance related consequences experienced.

CONTACTS AND LOCATIONS:
Overall Officials: Erin E Bonar, Ph.D., Principal Investigator — University of Michigan
Locations (1):
- Hurley Medical Center, Flint, Michigan, United States

IPD SHARING:
Plan to Share IPD: No